CLINICAL TRIAL: NCT01664676
Title: A Randomised, Double-blinded, Cross-over Study Investigating the Short-term Impact of Liraglutide on Kidney Function in Diabetic Patients
Brief Title: Effects of Liraglutide on Kidney Function in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Novo Nordisk A/S (Industry); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1131-5236; 2012-003577-26 (EudraCT Number)
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: liraglutide; victoza; GLP-1; kidney; diabetes; renal; diabetic nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Diabetic Nephropathies | interventions — Liraglutide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Experimental): 1.2 mg liraglutide sc. (single-dose)
  Interventions: Drug: Liraglutide
- Placebo-liraglutide (Placebo Comparator): Placebo liraglutide sc. (single-dose)
  Interventions: Drug: Placebo-liraglutide

INTERVENTIONS:
Drug: Liraglutide
  Other Names: Victoza
  Arms: Liraglutide
Drug: Placebo-liraglutide
  Other Names: Isotonic saline
  Arms: Placebo-liraglutide

SUMMARY:
Recent studies in rodents show that glucagon-like peptide-1 (GLP-1) analogues protect against diabetic nephropathy. We hypothesise that this is also the case in humans. This study will investigate the short-term effect of liraglutide (GLP-1 analogue) on the kidneys in type 2 diabetic patients. Impact on basic kidney physiological will be determined and kidney injury markers will be measured as surrogate parameters of kidney protection.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities.
* Male gender
* T2DM, diagnosed according to international guidelines
* Age 20-60 years, both included
* Body Mass Index (BMI): 20-32 kg/m2, both included
* Metformin treatment
* Albumin/creatinine ratio <25 mg/mmol

Exclusion Criteria:

* Known or suspected allergy to trial product or related products
* Previous participation in this trial
* Previous treatment with GLP-1 analogues or DPP-4 inhibitors
* Current treatment with any antidiabetic drug other than metformin
* Poorly regulated glycemic control (HbA1c > 8%)
* Impaired kidney function: estimated GFR < 70ml/min
* Impaired liver function: liver parameters exceed 2 times upper normal limit
* Subjects with active malignancy
* Severe cardiac insufficiency classified according to NYHA III-IV
* Unstable angina pectoris, acute myocardial infarction (AMI) within the last 12 months
* Severe, uncontrolled hypertension: sitting blood pressure (BP) > 180/110 mmHg
* Antihypertensive treatment consisting of more than two different pharmaceutical products
* Symptoms related to benign prostate hyperplasia
* Claustrophobia
* Any metal body implants
* History of pancreatitis, type 1 diabetes, gastroparesis or multiple endocrine neoplasia syndrome type 2
* Personal or family history of medullary thyroid carcinoma
* Any diseases judged by the investigator that could affect the trial
* Any medication judged by the investigator that could affect the trial

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Glomerular Filtration Rate (51Cr-EDTA plasma clearance) | 10-15 hours post-dose

SECONDARY OUTCOMES:
Renal Blood Flow (functional magnetic resonance imaging) | 15 hours post-dose
Renal electrolyte clearance | 10-15 hours post-dose
  Sodium, potassium, calcium, lithium and osmotically active substances.
Excretion of kidney injury markers | 0-10 hours and 10-15 hours post-dose
  Albumin, NGAL, KIM-1, angiotensinogen and 8-OHdG.
Plasma concentrations of various hormones | 10-15 hours post-dose
  Angiotensin II, renin, aldosterone, atrial natriuretic peptide, catecholamines.

CONTACTS AND LOCATIONS:
Overall Officials: Jens S Christiansen, Professor, Principal Investigator — Aarhus University Hospital, Department of Endocrinology and Diabetes
Locations (1):
- Aarhus University Hospital, Department of Endocrinology and Diabetes, Aarhus, Denmark